CLINICAL TRIAL: NCT03329742
Title: A Pilot Feasibility Study of Sipuleucel-T vs. Sipuleucel-T and Low-protein Diet in Patients With Metastatic Castrate-resistant Prostate Cancer (CRPC)
Brief Title: Sipuleucel-T and Low-protein Diet in Patients With Metastatic Castrate-resistant Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Nabil Adra, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0614; 1706081520 (Other: Indiana University IRB)
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer Recurrent
MeSH Terms: interventions — Diet, Protein-Restricted

STUDY DESIGN:
Intervention Model Description: This is a longitudinal randomized parallel groups design of n=30 subjects randomized in a 1:1 ratio to either sipuleucel-T plus control diet arm (20% protein content) or sipuleucel-T plus intervention low-protein content diet (10% protein diet).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control protein diet arm (Placebo Comparator): 20% protein content
  Interventions: Other: Control protein diet
- Low protein diet arm (Experimental): 10% protein content
  Interventions: Other: Low protein diet

INTERVENTIONS:
Other: Low protein diet — Patients on this arm will receive a prescribed diet (including all food and recommendations for beverages) that contains 10% protein to begin eating 1 week prior to treatment with sipuleucel-T and throughout treatment (i.e. diet will last approximately 49 days).
  Arms: Low protein diet arm
Other: Control protein diet — Patients on this arm will receive a prescribed diet (including all food and recommendations for beverages) that contains 20% protein to begin eating 1 week prior to treatment with sipuleucel-T and throughout treatment (i.e. diet will last approximately 49 days).
  Arms: Control protein diet arm

SUMMARY:
This is a single-center, randomized, open-label study to assess the feasibility of a low-protein diet intervention in patients with metastatic castrate-resistant prostate cancer (CRPC) who are receiving treatment with sipuleucel-T. Subjects will be randomized (1:1 ratio) to either Arm 1 or Arm 2 (Fig. 1).

Arm 1: Subjects randomized to Arm 1 will be treated with sipuleucel-T infusion on Day 1, every two weeks for a total of three infusions. Subjects on this arm will receive a control diet containing 20% protein.

Arm 2: Subjects randomized to Arm 2 will be treated with sipuleucel-T infusion on Day 1, every two weeks for a total of three infusions. Subjects on this arm will receive a low-protein diet containing 10% protein.

Patients with metastatic, asymptomatic or minimally symptomatic CRPC that has progressed despite androgen deprivation therapy will be eligible for the study. After informed consent eligible patients will be scheduled to receive sipuleucel-T (three infusions two weeks apart) with normal-protein diet vs. low-protein diet. Each cycle will be every 14 days. Diet intervention will commence 1 week prior to the first apheresis (Day -7) and will continue until 10 days after the last infusion of sipuleucel-T (Day +42) (Fig. 2).

DETAILED DESCRIPTION:
Primary Objective To assess the feasibility of low-protein diet intervention in patients with metastatic CRPC receiving immunotherapy with sipuleucel-T. Change in blood urea nitrogen (BUN) and urine urea nitrogen (UUN) from baseline to 6 weeks will be measured to assess adherence of following the diet intervention. The expected changes (mean, standard deviation) in BUN are 5.5 ± 2.6 mg/dL with 10% protein diet arm and 2.5 ± 2.6 mg/dL with 20% protein diet arm (please see section 12.5.7).

Secondary Objectives

1. To assess whether low-protein diet intervention augments the immune response to sipuleucel-T in men with metastatic CRPC.
2. To assess the safety and tolerability of the combination of sipuleucel-T and low-protein diet intervention.
3. To obtain preliminary evidence of clinical efficacy of the combination of sipuleucel-T and low-protein diet compared to sipuleucel-T and control-diet, including objective response rate (partial + complete response), progression-free survival (PFS) and overall survival (OS), and changes in prostate-specific antigen (PSA).

ELIGIBILITY:
ELIGIBILITY CRITERIA Men at least 18 years of age with asymptomatic or minimally symptomatic, metastatic, androgen independent prostate cancer will be recruited for this study. Before the initiation of screening procedures, the patient will undergo the Informed Consent Process which includes signing an Institutional Review Board (IRB)-approved consent form. The subject will subsequently undergo screening assessments to determine if he meets the eligibility criteria for the study.

Inclusion Criteria

* Histologically documented adenocarcinoma of the prostate.
* Metastatic disease as evidenced by soft tissue and/or bony metastases on baseline bone scan and/or computed tomography (CT) scan of the chest, abdomen, and pelvis
* Androgen independent prostatic adenocarcinoma. Subjects must have current or historical evidence of disease progression concomitant with surgical or medical castration, as demonstrated by PSA progression OR progression of measurable disease OR progression of non-measurable disease as defined below:

  * PSA: Two consecutive PSA values, at least 14 days apart, each ≥ 5.0 ng/mL and ≥ 50% above the minimum PSA observed during castration therapy or above the pre-treatment value if there was no response.
  * Measurable disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The change will be measured against the best response to castration therapy or against the pre-castration measurements if there was no response.
  * Non-measurable disease: Soft tissue disease: The appearance of 1 or more new lesions, and/or unequivocal worsening of non-measurable disease when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response.
  * Bone disease: Appearance of 2 or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response. Increased uptake of pre-existing lesions on bone scan does not constitute progression.
  * Serum PSA ≥ 5.0 ng/mL
  * Castration levels of testosterone (< 50 ng/dL) achieved via medical or surgical castration. Surgical castration must have occurred at least 3 months prior to registration. Subjects who are not surgically castrate must be receiving medical castration therapy, have initiated such therapy at least 3 months prior to registration, and continue such therapy until the time of confirmed objective disease progression.
* Life expectancy of at least 6 months
* Men ≥ 18 years of age
* Adequate hematologic, renal, and liver function as evidenced by the following:

  * White blood cell (WBC) ≥ 2,500 cells/μL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/μL
  * Platelet Count ≥ 100,000 cells/μL
  * Hemoglobin (HgB) ≥ 9.0 g/dL
  * Creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 2 x upper limit of normal (ULN)
  * Aspartate aminotransaminase (AST, SGOT) ≤ 2.5 x ULN
  * Alanine aminotransaminase (ALT, SGPT) ≤ 2.5 x ULN

Exclusion Criteria

* The presence of lung, liver, or known brain metastases, malignant pleural effusions, or malignant ascites.
* Moderate or severe symptomatic metastatic disease. Subjects who meet either of the following criteria must be excluded:

  * A requirement for treatment with opioid analgesics for any reason within 28 days prior to registration
  * Average weekly pain score of 4 or more as reported on the 10-point Visual Analog Scale (VAS) on the Registration Pain Log
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Use of non-steroidal antiandrogens (e.g., flutamide, nilutamide, or bicalutamide) within 6 weeks of registration.
* Treatment with chemotherapy within 28 days of registration including subjects who received more than 2 chemotherapy regimens in the metastatic setting at any time prior to registration.
* Treatment with any of the following medications or interventions within 28 days of registration:

  * Systemic corticosteroids; however, use of inhaled, intranasal, and topical steroids is acceptable.
  * Ketoconazole
  * High dose calcitriol [1,25(OH)2VitD] (i.e., > 7.0 μg/week)
  * Any other systemic therapy for prostate cancer (except for medical castration)
* Prior treatment with sipuleucel-T (on clinical trial or as part of standard of care)
* Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression
* Paget's disease of bone
* A history of stage III or greater cancer, excluding prostate cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer must have been adequately treated and been disease-free for ≥ 3 years at the time of registration.
* A requirement for systemic immunosuppressive therapy for any reason
* Any infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5°F or 38.1°C) within 1 week prior to registration
* A known allergy, intolerance, or medical contraindication to receiving the contrast dye required for the protocol-specified CT imaging
* Any medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for men with asymptomatic or minimally symptomatic, metastatic, androgen independent prostate cancer.
Enrollment: 2 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Adherence to diet intervention | 6 weeks
  BUN and UUN laboratory values

SECONDARY OUTCOMES:
Feasibility of diet intervention | 6 weeks
  Patient self-report of compliance
Feasibility of diet intervention | 6 weeks
  Rate of drop-out
Feasibility of diet intervention | 6 weeks
  Rate of enrollment
Safety and tolerability of diet intervention combined with sipuleucel-T treatment | 6 weeks
  Rate of adverse events per CTCAE
Rate of immune response | 6, 12, and 14 weeks
  IFN-γ ELISpot specific for PA2024 laboratory values
Progression free survival | 2 years
  Length of time during and after the treatment that a patient lives with the disease but it does not get worse
Overall survival | 2 years
  Length of time start of treatment that patients are still alive

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Adra, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No